CLINICAL TRIAL: NCT01373411
Title: Ticagrelor and Aspirin for the Prevention of Cardiovascular Events After Coronary Artery Bypass Surgery (CABG)
Brief Title: Ticagrelor and Aspirin for the Prevention of Cardiovascular Events After Coronary Artery Bypass Surgery
Acronym: TAP-CABG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cardiology Research UBC (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Dr. Jacqueline Saw, Principal Investigator, Cardiology Research UBC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H10-01452
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
Keywords: CABG; Ticagrelor; Coronary Artery Bypass Surgery
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo twice daily. Study drug will be started within 48 hours of CABG.
  Interventions: Drug: Placebo
- ticagrelor 90 mg (Active Comparator): Taken twice daily. Study drug will be started within 48 hours of CABG.
  Interventions: Drug: ticagrelor

INTERVENTIONS:
Drug: ticagrelor — ticagrelor 90 mg BID for 90 days
  Other Names: Brilinta
  Arms: ticagrelor 90 mg
Drug: Placebo — Placebo 1 pill BID for 90 days
  Arms: Placebo

SUMMARY:
Subjects will be consented to the study prior to Coronary Artery Bypass Graft (CABG) and randomly assigned to receive either ticagrelor 90 mg bid or placebo bid starting within 48 hours of surgery. Subjects will remain on study drug for a minimum of 12 months during which time they will receive telephone follow-up one and nine months following CABG and clinic visits three, six, and twelve months following CABG.

DETAILED DESCRIPTION:
Patients will be screened for eligibility pre-CABG, and informed consent signed before randomization. Aspirin 81mg/d will be started within 12 hours of CABG as per routine practice. Study medication will be started within 48 hours after CABG if there are no contraindications. Patients will be randomized to ticagrelor 90mg bid (no loading dose) or placebo bid for 1 year following CABG. Aspirin 81mg/d will be continued for at least 1 year post-CABG. Other cardiac medications will be at the discretion of the treating physicians as per standard practice.

Patients will be followed daily during their hospital stay. Outpatient visits will be scheduled at 3, 6 and 12 months. There will also be telephone contacts at 1 and 9 months.

CT Substudy:Patients in the CT angiography substudy(the first 240 enrolled subjects) will have a cardiac CT angiogram to evaluate bypass graft patency at 3-month follow-up.Grafts will be separately evaluated based upon the conduits used, internal mammary, radial, or saphenous vein grafts. Graft patency is defined as contrast filling of the conduit and the coronary artery beyond the anastomosis. Grafts with ≥50% stenosis will also be recorded. The location of the stenosis will also be recorded (proximal anastomosis, body of graft, or distal anastomosis). CT angiograms will be evaluated by 2 interpreters (radiologists or cardiologists) blinded to the randomized treatment, and will be reviewed by a 3rd interpreter if there are disagreements. If no consensus could be reached among the 3 interpreters, the graft will be deemed not analyzable, or be subject to invasive coronary angiography for definitive assessment if clinically indicated.

The primary efficacy endpoint is the composite of all-cause mortality, MI, stroke, or repeat revascularization within 1 year following CABG. Secondary endpoints include the individual endpoints of all-cause mortality, cardiovascular death, MI, stroke, repeat revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 19 years and ≤ 80 years old undergoing isolated CABG
2. Females of child-bearing age must have a negative pregnancy test at enrollment

Exclusion Criteria:

1. Patients undergoing combined valve or aortic surgeries
2. Patients requiring oral anticoagulant therapy on discharge that cannot be stopped (e.g. atrial fibrillation with CHADS2 score ≥ 2, pulmonary embolism, deep venous thrombosis)
3. Known allergy or intolerance to aspirin, clopidogrel or ticagrelor
4. Patients with active bleeding or history of bleeding diathesis
5. Patients with previous intracranial hemorrhage at any time, or ischemic stroke within 14 days
6. Patients with severe liver disease (e.g. ascites or signs of coagulopathy)
7. Patients with pre-operative or persistent post-operative Type 2 second-degree AV block, or 3rd degree AV block, without a permanent pacemaker
8. Patients with end-stage renal failure requiring dialysis
9. For patients enrolled in the CT angiography substudy, renal dysfunction with eGFR < 50 ml/min is an exclusion criteria

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality, MI, stroke, or repeat revascularization | within one year following CABG

SECONDARY OUTCOMES:
Improving graft patency | 3 months post-CABG
  The secondary study objective is to evaluate if the combination of ticagrelor and aspirin administered after CABG will improve graft patency at 3 months, compared with aspirin alone. This will be monitored and assessing in the CT angiography substudy.

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Saw, BSc, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Saw J, Wong GC, Mayo J, Bernstein V, Mancini GB, Ye J, Skarsgard P, Starovoytov A, Cairns J. Ticagrelor and aspirin for the prevention of cardiovascular events after coronary artery bypass graft surgery. Heart. 2016 May 15;102(10):763-9. doi: 10.1136/heartjnl-2015-308691. Epub 2016 Feb 18. PMID 26891756